CLINICAL TRIAL: NCT06864247
Title: Evaluating the Impact of Psoas Muscle Size, Composition, and Clinical Frailty on Long-term Outcomes Following Elective Endovascular Aneurysm Repair: a Multicenter Retrospective Study
Brief Title: Evaluating the Impact of Psoas Muscle Size, Composition, and Clinical Frailty on Long-term Outcomes Following Elective Endovascular Aneurysm Repair
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202407056RIND
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2024-08

CONDITIONS: Endovascular Aneurysm Repair (EVAR)
Keywords: Endovascular Aneurysm Repair (EVAR); Sarcopenia; Myosteatosis; Frailty
MeSH Terms: conditions — Sarcopenia; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The AAA patients undergoing EVAR procedures
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No intervention

SUMMARY:
Sarcopenia, which is characterized by the progressive loss of skeletal muscle mass and strength, has emerged as a significant prognostic biomarker in the field of vascular surgery, particularly regarding endovascular aneurysm repair (EVAR). This article delves into the implications of sarcopenia on the outcomes of EVAR, emphasizing its predictive value for long-term survival and potential as a tool for patient risk stratification.

Recent research suggests that sarcopenia could be used as a biomarker for prognosis. A systematic review and meta-analysis have underscored sarcopenia's negative prognostic value for survival during long-term follow-up post-EVAR. The presence of sarcopenia, as determined by decreased core muscle area in axial abdominal computed tomography (CT) scans, has been widely discussed as a predictor of outcomes in patients undergoing EVAR.1

Moreover, studies have consistently reported an association between sarcopenia and increased mortality and adverse outcomes following EVAR.2 For instance, a retrospective review investigating sarcopenia as a method to predict 1-year survival in patients undergoing EVAR found a significant increase in overall mortality among patients with the lowest quartile of normalized total psoas cross-sectional area (nTPA).2 Therefore, researchers suggested that physicians can use sarcopenia for risk stratification and patient selection before an EVAR. The evaluation of sarcopenia from preoperative CT scans can assist clinicians in identifying EVAR candidates who may be less likely to benefit from the procedure.2 This objective radiographic finding offers a standardized method for patient selection, which could be particularly useful in telemedicine and remote patient evaluation.

The integration of sarcopenia assessment into the preoperative evaluation of patients considered for EVAR can revolutionize the approach to managing abdominal aortic aneurysms (AAA). By providing a reliable biomarker for risk stratification, sarcopenia can enable a more personalized treatment plan, potentially improving patient outcomes and optimizing healthcare resources. Nonetheless, the majority of the studies were conducted among Western populations. The implications are questionable for Taiwan patients. This study aims to fill the gap and to analyze the sarcopenia and its impact on patient outcomes following EVAR in Taiwan

ELIGIBILITY:
Inclusion Criteria:

* The AAA patients undergoing EVAR procedures

Exclusion Criteria:

* The AAA patients undergoing open surgery procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The AAA patients undergoing EVAR procedures
Sampling Method: Probability Sample
Enrollment: 525 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-01-03 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
Death | From enrollment to the end at 8 years
  The social security death was queried to confirm all deaths and survey patients lost to follow-ups

SECONDARY OUTCOMES:
Clinical outcomes | From enrollment to the end at 8 years
  Clinical adverse events, number of participants with cardiac events, number of participants with cerebrovascular events, number of participants with amputation events, number of participants with accesssite events, number of participants with reintervention events.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided